CLINICAL TRIAL: NCT07266935
Title: A Prospective, Randomized Controlled Trial Evaluating the Effectiveness of Posterior Pericardiotomy in Preventing Postoperative Atrial Fibrillation Among Yemeni Cardiac Surgical Patients
Brief Title: Posterior Pericardiotomy for Prevention of POAF After Cardiac Surgery: RCT in Yemen
Acronym: PP-POAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taiz University - Faculty of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TaizU-PP-AF-2022
Record Dates: First submitted 2025-09-26; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Atrial Fibrillation; Cardiac Tamponade
Keywords: Posterior pericardiotomy; Postoperative atrial fibrillation; Cardiac tamponade; Yemen
MeSH Terms: conditions — Cardiac Tamponade | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors were blinded to the treatment group; participants and care providers were aware of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional: Posterior Pericardiotomy (Experimental): A longitudinal posterior pericardiotomy incision (4-5 cm) is made parallel and posterior to the left phrenic nerve during open-heart surgery. This intervention aims to reduce postoperative atrial fibrillation, pericardial effusion, and cardiac tamponade.
  Interventions: Procedure: Posterior Pericardiotomy
- Control: Standard Care (Active Comparator): Conventional open-heart surgery is performed without posterior pericardiotomy. Standard perioperative care is provided.
  Interventions: Procedure: Standard Care

INTERVENTIONS:
Procedure: Posterior Pericardiotomy — A longitudinal posterior pericardiotomy incision (4-5 cm) is made parallel and posterior to the left phrenic nerve during open-heart surgery.
  Arms: Interventional: Posterior Pericardiotomy
Procedure: Standard Care — Conventional open-heart surgery without posterior pericardiotomy. Standard perioperative care is provided.
  Arms: Control: Standard Care

SUMMARY:
A single-center, randomized controlled trial in Yemen evaluating whether posterior pericardiotomy (PP) reduces postoperative atrial fibrillation (POAF) after open-heart surgery. 210 patients undergoing CABG, aortic valve replacement, ascending aortic surgery, or combined procedures were randomized 1:1 to receive either posterior pericardiotomy (PP group, n = 106) or standard care (control group, n = 104). Outcomes assessed included POAF incidence, pericardial effusion, cardiac tamponade, ICU stay, mechanical ventilation, in-hospital mortality, and re-exploration for bleeding or tamponade.

DETAILED DESCRIPTION:
This single-center, prospective randomized controlled trial was conducted at the Cardiovascular and Kidney Transplantation Centre, Taiz University, Yemen. Adult patients undergoing elective open-heart surgery were randomized to receive either posterior pericardiotomy or standard care. The intervention involved creating a longitudinal posterior pericardiotomy incision parallel to the left phrenic nerve to facilitate pericardial drainage into the left pleural cavity.

The study evaluated the impact of posterior pericardiotomy on postoperative atrial fibrillation and related complications, including pericardial effusion and cardiac tamponade, compared with standard surgical management. Participants were monitored during hospitalization and followed for 30 days after surgery to assess clinical outcomes, resource utilization, and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Elective open-heart surgery:

Coronary artery bypass grafting (CABG) Aortic valve replacement Ascending aortic surgery Combined procedures (e.g., CABG + valve replacement)

Exclusion Criteria:

* Previous cardiac or thoracic surgery
* Left-sided pleural adhesions
* Preoperative atrial fibrillation or other rhythm disorders
* Hyperthyroidism
* Renal failure with plasma creatinine >2.0 mg/dL
* Off-pump CABG
* Mitral or tricuspid valve surgery (excluded due to distinct pathophysiology and POAF risk)
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative atrial fibrillation (POAF) until hospital discharge | During hospitalization, approximately 5-7 days
  Occurrence of atrial fibrillation documented by 12-lead ECG or continuous telemetry monitoring, lasting >30 seconds, and occurring after cardiac surgery in patients with no prior history of atrial fibrillation.

SECONDARY OUTCOMES:
Number of participants requiring postoperative antiarrhythmic medications | From surgery until hospital discharge (average 7-10 days)
  Any antiarrhythmic therapy administered postoperatively to manage POAF
Number of Participants Requiring Systemic Anticoagulation or Cardioversion for Arrhythmia | From surgery until hospital discharge (average 7-10 days)
  Any anticoagulation therapy or cardioversion performed for arrhythmia management
Number of participants with cardiac tamponade requiring intervention | From date of surgery through 30 days postoperatively
  Clinically diagnosed cardiac tamponade requiring intervention
Number of participants requiring surgical re-exploration for bleeding or tamponade | From date of surgery through 30 days postoperatively
  Any return to surgery for bleeding or tamponade relief
Duration of Mechanical Ventilation (Hours) | From end of surgery until successful extubation (up to 72 hours postoperatively)
  Total hours under mechanical ventilation until successful extubation
Duration of ICU stay (hours) | From ICU admission after surgery until transfer to ward (average of 1-4 days)
  Total time in ICU from admission to transfer to ward
Duration of total hospital stay (days) | From date of surgery until hospital discharge (average of 7-10 days)
  Days from surgery to discharge
Number of participants with in-hospital mortality (any cause) | From date of surgery until hospital discharge (average of 7-10 days)
  Death from any cause during hospital stay
Number of participants experiencing major adverse cardiovascular events (MACE: stroke, myocardial infarction, or death) | From date of surgery through 30 days postoperatively
  Occurrence of stroke, myocardial infarction, or all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ismail S Al Shameri, MD, Principal Investigator — Cardiovascular & Kidney Transplantation Centre, Taiz University, Yemen
Locations (1):
- Cardiovascular & Kidney Transplantation Centre, Taiz University, Taiz, Yemen, Taiz, Muḩāfaz̧at Ta‘izz, Yemen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Shameri I, Al-Ganadi AA, Noman T, Kadry MA, Elsharkawy IM, Al-Wsabi N, Mohammed AA. Posterior Pericardiotomy and Its Impact on Cardiac Tamponade and Pericardial Effusion after Cardiac Surgery. Ann Thorac Cardiovasc Surg. 2025;31(1):25-00075. doi: 10.5761/atcs.oa.25-00075. PMID 40603058